CLINICAL TRIAL: NCT03152123
Title: A Randomized, Double-Blind, Active- and Placebo-Controlled, Single-Dummy, 4-Way Crossover Study to Determine the Abuse Potential of Pitolisant Compared to Phentermine and Placebo, in Healthy, Non-Dependent Recreational Stimulant Users
Brief Title: Determination the Abuse Potential of Pitolisant in Healthy, Non-Dependent Recreational Stimulant Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioprojet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P16-02 / BF2.649
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Healthy; Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — pitolisant; Phentermine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pitolisant HCl, 40 mg (Experimental): Pitolisant HCl, 40 mg administered as 2 capsules, each containing 1 × 20 mg pitolisant HCl tablet (over-encapsulated), and 2 capsules, each containing 1 × 100 mg lactose tablet (over-encapsulated)
  Interventions: Drug: Pitolisant
- Pitolisant HCl, 240 mg (Experimental): Pitolisant HCl, 240 mg administered as 4 capsules, each containing 60 mg pitolisant HCl (3 x 20 mg pitolisant HCl tablets, encapsulated in 1 capsule)
  Interventions: Drug: Pitolisant
- Phentermine HCl, 60 mg (Active Comparator): Phentermine HCl, 60 mg administered as 2 capsules, each containing 1 × 30 mg phentermine HCl capsule (over- encapsulated), and 2 capsules, each containing 1 × 100 mg lactose tablet (over-encapsulated)
  Interventions: Drug: Phentermine
- Placebo (Placebo Comparator): Placebo administered as 4 capsules, each containing 1 × 100 mg lactose tablet (over-encapsulated)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Pitolisant — Pitolisant 40 mg or 240 mg (tablets over-capsuled)
  Other Names: BF2.649
  Arms: Pitolisant HCl, 240 mg; Pitolisant HCl, 40 mg
Drug: Placebos — tablets over-capsuled
  Arms: Placebo
Drug: Phentermine — Phentermine 60 mg (capsule over-capsuled)
  Arms: Phentermine HCl, 60 mg

SUMMARY:
The purpose of this study is to assess the abuse potential of single doses of pitolisant relative to phentermine HCl and placebo, when administered to healthy, non-dependent, recreational stimulant users.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects 18 to 55 years of age, inclusive.
* Must understand and provide written informed consent, prior to the initiation of any protocol-specific procedures.
* Current stimulant users who have used stimulants for recreational (non-therapeutic) purposes, (ie, for psychoactive effects) at least 10 times in the past year and used stimulants at least 1 time in the 8 weeks before Screening.
* Female subjects of childbearing potential with male sexual partners must be using and willing to continue using medically acceptable contraception for at least 1 month prior to Screening (at least 3 months for oral and transdermal contraceptives) and for at least 1 month after last study drug administration.
* Male subjects with female sexual partners of childbearing potential must be using and willing to continue using medically acceptable contraception from Screening and for at least 1 month after the last study drug administration.
* Able to speak, read, and understand English sufficiently to allow completion of all study assessments.

Exclusion Criteria:

* Substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition - Text Revision (DSM IV-TR), and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
* History or presence of clinically significant abnormality as assessed by physical examination, medical history, vital signs, or laboratory values, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results.
* History or presence of motor tics, Tourette's syndrome, or significant anxiety, tension, or agitation.
* Presence of thyrotoxicosis, advanced arteriosclerosis, glaucoma, pheochromocytoma, acid related gastric disorders, or peripheral vasculopathy (including Raynaud's phenomenon).
* History or presence of cardiovascular disorder (eg, moderate to severe hypertension, angina, arterial occlusive disease, heart failure, hemodynamically significant congenital heart disease, cardiomyopathies, myocardial infarction, potentially life-threatening arrhythmias and channelopathies [disorders caused by the dysfunction of ion channels]), or other serious cardia problems.
* History or presence of CNS abnormalities (eg, cerebral aneurysm, vascular abnormalities, stroke), seizures, convulsions, or epilepsy.
* History or presence of clinically significant abnormality as assessed by ECG, long QTc syndrome (eg, syncope or arrhythmia), or presence QTcF interval >450 msec.
* Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase or aspartate aminotransferase > 1.5 × the upper limit of normal (ULN) or bilirubin > 1 × ULN.
* Positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* History of allergy or hypersensitivity to pitolisant, phentermine HCl, or related drugs (eg, sympathomimetic amines) or known excipients of any of the drug products in this study (eg, lactose).
* History of severe allergic reaction (including anaphylaxis) to any substance or previous status asthmaticus.
* Subjects with any history of suicidal ideation or suicidal behavior, as assessed by the C SSRS (baseline version).
* Treatment with an investigational drug within 5 times the elimination half-life, if known (eg, a marketed product), or within 30 days (if the elimination half-life is unknown) prior to the first study drug administration or is concurrently enrolled in any research, judged not to be scientifically or medically compatible with this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Maximum effect (Emax) on Drug Liking visual analog scale (VAS) | Within 24 hours post-dose
  Drug liking VAS is one of the measures of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm).

SECONDARY OUTCOMES:
Drug Liking VAS (minimum effect [Emin] and time-averaged area under the effect curve to 24 hours after study drug administration [TA_AUE]) | Within 24 hours post-dose
  Drug liking VAS is one of the measures of balance of effects that assesses the degree that a participant likes a drug effect at the time the question is being asked (that is, at the moment). It is scored using a 100 millimeter (mm) bipolar visual analogue scale (VAS) anchored in the center with a neutral anchor of "neither like nor dislike" (score of 50 mm), on the left with "strong disliking" (score of 0 mm) and on the right with "strong liking" (score of 100 mm).
Overall Drug Liking VAS (Emax/Emin) | Within 24 hours post-dose
  Overall drug liking VAS is one of the measures of balance of effects that assesses the participant's global perception of drug liking (that is, effects over the whole course of the drug experience including any carryover effects). A 100 mm bipolar VAS is used to assess response based on a score ranging from 0 mm to 100 mm (0 mm = "strong disliking", 50 mm= "neither like nor dislike", and 100 mm= "strong liking").
Take Drug Again VAS (Emax) | Within 24 hours post-dose
  Take drug again VAS is one of the measures of balance of effects. It is a subjective assessment of the degree to which a participant would desire to take the drug again if given the opportunity. It is presented on a 100 mm bipolar VAS with score ranging from 0 mm to 100 mm (score of 0 mm = "definitely not", 50 mm = "do not care", and 100 mm = "definitely so").
Good Effects VAS (Emax and TA_AUE) | Within 24 hours post-dose
  Good drug effects VAS is one of the measures of positive effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
Bad Effects VAS (Emax and TA_AUE) | Within 24 hours post-dose
  Bad effects VAS is one of the measures of negative effects that assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= definitely not) to 'extremely' (score of 100 mm= definitely so).
ARCI-A scale (Emax and TA_AUE) | Within 24 hours post-dose
  ARCI-A is measure of other stimulant effects. It is a set of 13 questions in which each question contributes to total score. Participants select 'False' / 'True' for response. One point given for each response that agrees with scoring direction, true items receive score of 1 if answer 'True', false items receive score of 1 if answer 'False'. No points if answer is opposite to scoring direction. Score range: 0 to 13, higher score indicated higher other subjective effects.
ARCI-BG scale (Emax and TA_AUE) | Within 24 hours post-dose
  ARCI-BG is measure of other subjective effects. It is a set of 13 questions in which each question contributes to total score. Participants select 'False' / 'True' for response. One point given for each response that agrees with scoring direction, true items receive score of 1 if answer 'True', false items receive score of 1 if answer 'False'. No points if answer is opposite to scoring direction. Score range: 0 to 13, higher score indicated higher other subjective effects.
Agitation/Relaxation VAS (Emax and TA_AUE) | Within 24 hours post-dose
  Agitation/Relaxation VAS assesses the effect experienced by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm) to 'extremely' (score of 100 mm).
Drug Similarity VAS (score at 24 hours after study drug administration) | Within 24 hours post-dose
  Drug similarity VAS is one of the measures of other subjective effects. It assesses the similarity of the drug recently received by the participant on a 100 mm unipolar VAS, where responses are unidirectional and range from a response of 'none' (score of 0 mm= not at all similar) to 'extremely' (score of 100 mm= very similar).
Safety and tolerability of Pitolisan HCl as assessed by AEs | Up to 6 weeks
  AEs assessment
Safety and tolerability of Pitolisan HCl by laboratory assessments | Up to 6 weeks
  Laboratory assessments
Safety and tolerability of Pitolisan HCl as assessed by 12-lead ECGs | Up to 6 weeks
  12-lead ECGs assessments
Safety and tolerability of Pitolisan HCl as assessed by vital signs | Up to 6 weeks
  Vital signs assessment
Safety and tolerability of Pitolisan HCl as assessed by physical examination | Up to 6 weeks
  Physical examination assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael B. McDonnell, MD, Principal Investigator — Syneos Health
Locations (1):
- INC Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Setnik B, McDonnell M, Mills C, Scart-Gres C, Robert P, Dayno JM, Schwartz JC. Evaluation of the abuse potential of pitolisant, a selective H3-receptor antagonist/inverse agonist, for the treatment of adult patients with narcolepsy with or without cataplexy. Sleep. 2020 Apr 15;43(4):zsz252. doi: 10.1093/sleep/zsz252. PMID 31626696